CLINICAL TRIAL: NCT05237739
Title: Clinical- and Patient-reported Outcomes Following Treatment of Grade III Furcation-involved Molars. A Single-centre Single-masked Randomised Controlled Feasibility Trial With SMART Design.
Brief Title: Treatment of Advanced Grade III Periodontal Furcation Lesions
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23012022
Record Dates: First submitted 2022-01-24; First posted 2022-02-14 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Furcation Defects; Periodontitis; Surgical Procedure, Unspecified; Periodontal Bone Loss
MeSH Terms: conditions — Furcation Defects; Periodontitis; Alveolar Bone Loss

STUDY DESIGN:
Intervention Model Description: This is a single-centre single-masked randomised controlled feasibility trial with SMART design to assess the response to treatment for degree III periodontal furcation involved molars (n=20).
Who Masked: Investigator, Outcomes Assessor
Masking Description: Simple randomisation will be completed using the online programme, Sealed Envelope. This will be completed by a member of the research team not involved in this specific study. Sealed Envelope will provide a randomisation schedule, patient numbering and a sequence of patient number assignment. This will all be safely stored and secured. The treatment allocation will be communicated to the study therapist/nurse and patient when booking the treatment appointment. It will not be possible to blind the participants or the clinician completing the study treatment. The study examiner will remain blind to treatment allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): Ten participants will be randomised to receive surgical periodontal treatment in the form of open flap debridement (OFD).
  Interventions: Procedure: Open Flap Debridement (OFD)
- Control Group (Active Comparator): Ten participants will be randomised to receive non-surgical periodontal treatment (NSPT). All treatment will be carried out by the same therapist, including oral hygiene.
  Interventions: Procedure: Non-Surgical Periodontal treatment (NSPT)

INTERVENTIONS:
Procedure: Non-Surgical Periodontal treatment (NSPT) — Participants will receive local anesthesia. Thorough debridement of the root surface will be completed to the depth of the periodontal pocket and of the furcation lesion, by using piezo-electric/ultrasonic devices with specific thin and delicate tips (such as Cavitron, Dentsply Sirona, US) and/or curettes. Treatment chair time will be recorded for each visit.
  Arms: Control Group
Procedure: Open Flap Debridement (OFD) — Patients will receive local anesthesia and intrasulcular incisions will be made by buccal and lingual/palatal aspects in order to reflect full-thickness flaps. After reflection of the flaps, the granulation tissue around the tooth will be removed with the non-cutting edge of a suitable scaling instrument such as a curette, taking care not to damage the root surfaces. Thorough debridement of the furcation area will be carried out by using piezo-electric/ultrasonic devices with specific thin and delicate tips
  Arms: Test Group

SUMMARY:
Periodontitis, a microbially-driven inflammatory disease has been shown to be the sixth most common disease of mankind. The 2009 UK Adult Dental Health Survey found that 54% of adults experience gum bleeding (gingivitis) with 45% of these suffering from periodontitis. Periodontitis begins at the gingival margins of teeth and over time, in susceptible individuals, the presence of a plaque biofilm can lead to the loss of the supporting connective tissue and alveolar bone associated with the teeth. This leads to the formation of a pathological periodontal pocket between the gingiva and tooth root, measurable by the use of a periodontal probe and recorded as the probing pocket depth (PPD). The associated loss of alveolar bone support is measurable radiographically and often leads to tooth mobility and if allowed to persist, can eventually lead to tooth loss. Periodontitis is classified into 4 stages (I-IV) based on disease severity and 3 grades (A-B-C) based on risk of disease progression.

The treatment of periodontitis involves a non-specific reduction of the bacterial load below the gingival margin. This is achieved by effective oral hygiene procedures and non-surgical periodontal therapy (NSPT), both of which are aimed at the removal of calculus (tartar) deposits and the disruption of the plaque biofilm from the affected root surfaces. In some cases, this treatment may then be followed by more invasive treatments such as periodontal surgery and if successful, patients can then be followed and maintained with supportive periodontal maintenance therapy (SPT). It should be noted that certain periodontal lesions in some patients do not however always respond favourably to treatment.

DETAILED DESCRIPTION:
Study teeth will have received at least one course of non-surgical periodontal treatment (NSPT) prior inclusion to the trial. At the baseline appointment participants will be randomly assigned to a treatment arm to receive either non-surgical periodontal treatment (n=10) or surgical periodontal treatment (n=10) for the first treatment phase. This is consistent with standard periodontal treatment procedures as it has been shown that either treatment can be considered as a valid option for cases of periodontitis where residual periodontal pocketing remains.

Simple randomisation will be completed using the online programme, Sealed Envelope. This will be completed by a member of the research team not involved in this specific study. Sealed Envelope will provide a randomisation schedule, patient numbering and a sequence of patient number assignment. This will all be safely stored and secured. The treatment allocation will be communicated to the study therapist/nurse and patient when booking the treatment appointment. It will not be possible to blind the participants or the clinician completing the study treatment. The study examiner will remain blind to treatment allocation.

For treatment stage II (after the 6-month evaluation), only 'non-responders' will be randomised further. Two new randomisation sequences (one for the initial non-surgical arm and one for the initial surgical arm) will be generated by Sealed Envelope for this purpose. If all participants in one treatment group are deemed non-responsive, the maximum number of participants randomised to each treatment arm in treatment stage II will be 5 (assuming no drop-outs or participants lost to follow up).

Non-Surgical Periodontal treatment (NSPT)

Ten participants will be randomised to receive non-surgical periodontal treatment (NSPT). All treatment will be carried out by the same therapist, including oral hygiene. The protocol for NSPT is as follows:

Participants will receive local anesthesia. Thorough debridement of the root surface will be completed to the depth of the periodontal pocket and of the furcation lesion, by using piezo-electric/ultrasonic devices with specific thin and delicate tips (such as Cavitron, Dentsply Sirona, US) and/or curettes. Treatment chair time will be recorded for each visit.

Open Flap Debridement (OFD)

Ten participants will be randomised to receive surgical periodontal treatment in the form of open flap debridement (OFD). The protocol for this procedure is based as follows:

Patients will receive local anesthesia and intrasulcular incisions will be made by buccal and lingual/palatal aspects in order to reflect full-thickness flaps. After reflection of the flaps, the granulation tissue around the tooth will be removed with the non-cutting edge of a suitable scaling instrument such as a curette, taking care not to damage the root surfaces. Thorough debridement of the furcation area will be carried out by using piezo-electric/ultrasonic devices with specific thin and delicate tips (such as Cavitron, Dentsply Sirona, US) and/or curettes. No ostectomy (excision of a portion of bone) will be completed, but osteoplasty (reshaping/removal of non-supporting bone) may be carried out, as judged by the operator. The surgical site will be closed with resorbable sutures. Participants will be given detailed post-operative instructions regarding care for the site after surgery and they will return one week later for removal of the sutures and a review of the surgical site. Treatment time will be completed for each visit.

Reassessment and definition of 'responsive to treatment' This clinical trial is based on the principles of a SMART designed trial. As part of this proposal, 20 participants will be randomised to receive either surgical or non-surgical treatment of teeth with furcation lesions, this will be known as the treatment I phase. At the 6 months post baseline reassessment (visit 6), 'response' will be assessed. Participants will be deemed 'responsive to treatment' or 'non-responsive to treatment' depending on a combination of clinical and patient-reported parameters Following the initial 6-month reassessment and in line with the principles of a SMART trial, the treatment for each patient, i.e. treatment phase II, will be either 'augmented', 'continued' or 'stepped down'. This second phase of treatment will be a logical, sequential continuation of treatment following on from treatment phase I. The options available to each participant will be dependent upon the treatment arm to which the participant was first randomised (surgical or non-surgical treatment) and their response to that specific treatment (i.e., responsive or non-responsive).

Non-surgical periodontal treatment (NSPT) with local antibiotics Local antimicrobials are often used as adjunctive therapy to subgingival debridement in the treatment of periodontitis. It has been suggested that when used in particular disease conditions, adjunctive local antimicrobials may be able to improve clinical outcomes.

NSPT will be carried out in the same fashion as described above. In addition to this, patients allocated to the local antibiotic group will receive local antibiotics (Dentomycin/ 2% minocycline) in the furcation area of the study tooth. The medication will be administered into the pocket with the applicator provided by the manufacturer to fill the pocket up to the gingival margin. Participants in the local antibiotics arm will be advised to avoid any form of interdental or inter-furcational cleaning (flossing, brushing, etc.) for the first 36 hours following treatment. After 36 hours normal oral hygiene procedures can be resumed. Treatment chair time will be recorded for each visit.

Saliva sampling All subjects should refrain from eating or drinking for at least 1 hour prior to saliva sampling. After a water rinse, donors will allow saliva to collect in their mouths before gently expectorating into a sterile 5 ml conical or other appropriate tube (alternatively to be pipetted to a 5 ml tube from a sterile bowl), which will then be placed on ice before being transferred to a laboratory freezer for storage at or below -70°C for storage and analysis at the end of the study.

Gingival crevicular fluid sampling The test site (TS) to be treated will undergo GCF sampling. A 'control site' (CS) will be chosen for sampling for each patient among buccal sites. The 'control' site will be a site with PPD<4mm and not bleeding on probing at the screening visit (if available a molar comparison site without furcation involvement will be chosen as a control for furcation sites). Samples of GCF will be collected from the selected TS and CS at baseline and at the treatment 2, 1-month, 6-month and 12-month follow-ups, prior to periodontal probing to avoid contamination by blood. Saliva will be removed from the supra-gingival area using saliva ejector and cotton rolls, being careful not to touch the gingival margin area; supra-gingival plaque, if present, will be removed using a curette to prevent saliva and/or plaque contamination. GCF will be collected for 30 seconds using methylcellulose strips carefully placed gently at the entrance of the sulcus until slight resistance is felt. GCF volume will be measured by Periotron, after which GCF will be extracted in acidic buffer to better preserve inflammatory mediators of periodontal disease from breakdown and/or oxidative processes, which occur to a major extent on the paper strips during storage. GCF samples will be then placed into small conic vials and stored at between -70 and -80°C until time of analysis aimed at assessing inflammatory, oxidative stress and wound healing markers in GCF before and after treatment in test and control sites.

Subgingival plaque sampling Following GCF collection, the 'test site' (TS) will have samples of subgingival plaque collected from the palatal/lingual aspect. A 'control site' (CS) will be chosen for sampling for each patient among buccal sites. The CS will be a site with PPD<4mm and not bleeding on probing at the screening visit (if available a molar comparison site without furcation involvement will be chosen as a control for furcation sites). Plaque samples will be collected from the selected TS and CS at baseline, 6-month and 12-month follow-ups.

Ahead of the sampling procedure, the supra-gingival plaque will be carefully removed, the site isolated with cotton rolls and gently dried. A sterile curette will then be inserted into the bottom of the pocket and removed after a single stroke and the content will be placed in a test tube containing reduced transport fluid until time of analysis, aimed at assessing the composition of the subgingival microbiota before and after treatment in test and control sites.

End of Study Definition The study would be considered completed after 30 months after the last patient last visit and all pertinent analyses.

However, if some patients needed further treatment to stabilise the condition of their gums, this would be offered at the hospital at the discretion of the consultant in charge and it would not be part of the study.

ELIGIBILITY:
Inclusion Criteria:

The following criteria will be considered for inclusion in the study:

* Age 18-70
* Diagnosis of Periodontitis stage III or IV, grade A, B or C
* At least one maxillary or mandibular molars with:
* Furcation involvement grade III horizontal classification degree B-C vertical classification without any ongoing restorative problems as judged by the study clinician)
* Probing depth ≥ 6mm
* Mobility < degree II (as examined by the study clinician)
* Absence of any ongoing endodontic pathology (as examined by the study clinician)
* Absence of an adjacent tooth with unfavorable periodontal prognosis (as judged by the study clinician)
* Non-surgical periodontal therapy performed to the study site within the last 6 months.
* Able to consent to study participation

Exclusion Criteria

* Smoking (any current or in past 5 years)
* Medical history including diabetes or hepatic or renal disease, or other serious medical conditions or transmittable diseases
* History of conditions requiring prophylactic antibiotic coverage prior to invasive dental procedures
* Anti-inflammatory or anticoagulant therapy during the month preceding the baseline exam
* Systemic antibiotic therapy during the 3 months preceding the baseline exam
* History of alcohol or drug abuse

  •. Self-reported pregnancy or lactation
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that according to the investigator may increase the risk associated with trial participation
* Previous surgical periodontal performed to the study site.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-02-05 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Number of patients | 13 months
  Number of participants recruited and retained into the study
Number of responsive and non-responsive | 13 months
  Number of participants deemed responsive and non-responsive to different treatments. Questionnaire will be used to assess the responsiveness to each treatment.
Number of participants randomised | 13 months
  Number of participants willing to be randomised to treatment II of the study (if deemed non-responsive following treatment I). Yes or Not answer to randomisation will be used to assess this number.
patient-reported outcomes (Pros) | 13 months
  A self-administered questionnaire will be used to assess the patient-reported outcomes (PROS) at 6 and 12 months based on different treatment arms
Probing Pocket Depth (PPD) | 13 months
  Distance between gingival margin and the bottom of the pocket, measured in mm
Bleeding on probing (BOP) | 13 months
  Bleeding after probing with the periodontal probe the gingival margin, 0 no bleeding 1 bleeding.

SECONDARY OUTCOMES:
Microbiological analysis | 13 months
  Sub gingival plaque will be collected from each participant and after DNA extraction a shot-gun metagenomic analysis will be used. This technique sequences DNA from many cultured microorganisms and the human genome. Randomly shears DNA will reconstructs into a consensus sequence. Shotgun sequencing reveals genes present in environmental samples with advances in high throughput sequencing technologies. Shotgun metagenomics provides information both about which organisms are present and what metabolic processes are possible in the community. Our aim is to assess which processes are possible in the community.

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Nibali, Principal Investigator — Floor 18, Tower Wing Guy's Hospital London SE1 9RTN/A
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No